CLINICAL TRIAL: NCT07031635
Title: The Effect of Hydrotherapy During Labor on Labor Pain, Duration of Labor, Birth Affectivity, and Breastfeeding
Brief Title: Hydrotherapy in Labor: Outcomes for Pain, Birth, and Breastfeeding
Acronym: HYDROTHERAPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Hacer ALAN DİKMEN, Assoc. Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/1177
Record Dates: First submitted 2025-06-03; First posted 2025-06-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy; Latent Phase
Keywords: Breast Feeding; Labor; Hydrotherapy; Labor Pain
MeSH Terms: conditions — Breast Feeding; Labor Pain | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: Randomized control study:
  The pilot study was conducted between July 16 and August 15, 2024, with 10 primiparous pregnant women. Hydrotherapy was applied and the usability of data collection forms was assessed. Participants were satisfied with the application, and no revisions to the forms were needed.
  Intervention Group:
  When cervical dilation reached 5 cm, participants received a 30-minute warm shower, either standing or sitting based on their preference. Various assessment tools were used throughout labor, including the Visual Analog Scale, Labor Monitoring Form, LATCH Breastfeeding Scale, and Labor Affect Scale.
  Control Group:
  Aside from routine hospital procedures, no additional interventions were performed. The same assessment tools were applied during labor and postpartum.
Who Masked: Participant, Outcomes Assessor
Masking Description: To prevent bias in the study sample, inclusion, exclusion, and withdrawal criteria were established.
  The intervention was performed solely by the researcher, therefore performance bias could not be prevented.
  Group assignments were done using random numbers generated by random.org, placed in opaque sealed envelopes, and assigned by an independent person not involved in the study. This ensured that participants were blinded to their group allocation.
  All data were collected by the researcher, who was aware of the group assignments; thus, measurement bias could not be prevented. However, data analyses were conducted by an independent statistician not involved in the research process, preventing statistical bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HYDROTHERAPY Group (Experimental): Pregnant women who met the inclusion criteria and agreed to participate in the intervention group received a warm shower once cervical dilation reached 5 cm. Based on their preference, participants either stood or sat during the 30-minute shower. After random assignment, the participants in the intervention group completed the "Informed Consent Form," "Personal Information Form," and the "Visual Analog Scale (VAS)" upon admission to the delivery room. During the 1st, 2nd, 3rd, and 4th stages of labor, the "Labor Monitoring Form" was used, and the VAS was repeated immediately after the intervention, and again at 30 and 60 minutes. Breastfeeding status was assessed using the LATCH scale within the first two hours after birth, and emotional responses to birth were evaluated using the Labor Affect Scale.
  Interventions: Other: Hydrotherapy (Warm Shower)
- Control group (No Intervention): In the control group, routine hospital procedures were followed, including admission, history-taking, informed consent, recording of vital signs, and connecting the mother to the non-stress test (NST) monitor. No additional intervention was administered. After random assignment, control group participants also completed the "Informed Consent Form," "Personal Information Form," and "Visual Analog Scale" at admission. The "Labor and Postpartum Monitoring Form" was used during the 1st through 4th stages of labor, and the VAS was repeated at 30 and 60 minutes after entering the active phase. Within the first two hours postpartum, breastfeeding was evaluated using the LATCH scale, and emotional responses to birth were assessed using the Labor Affect Scale.

INTERVENTIONS:
Other: Hydrotherapy (Warm Shower) — Pregnant women who met the inclusion criteria and agreed to participate in the intervention group received a warm shower once cervical dilation reached 5 cm. Based on their preference, participants either stood or sat during the 30-minute shower.
  Arms: HYDROTHERAPY Group

SUMMARY:
Warm showers are increasingly gaining attention for their positive impact on labor, yet studies on this topic in Turkey remain limited. No previous research has simultaneously evaluated the effects of warm showers on labor pain, duration, emotional state, and breastfeeding. As a simple, economical, accessible, and side-effect-free method, warm showers represent a practical and safe non-pharmacological option for pain relief and comfort during labor. This study aimed to evaluate the effects of hydrotherapy on labor pain, duration, breastfeeding, and emotional experience during childbirth.

DETAILED DESCRIPTION:
Childbirth is an unforgettable and unique experience for women. However, labor can sometimes be painful, challenging, and anxiety-inducing. Severe labor pain can negatively affect a woman's sense of control during labor, causing stress that may impact the health of the mother, fetus, and newborn. Traumatic birth experiences may hinder maternal-infant bonding and breastfeeding. Factors such as delivery method, medical interventions, pain, and fatigue can delay the initiation of breastfeeding and complicate the mother's adjustment to her new role. In supportive, intervention-free birth environments, the need for analgesia and oxytocin is reduced, episiotomy rates are lower, maternal emotional experiences improve, and breastfeeding is initiated earlier.

In this context, non-pharmacological methods such as warm showers offer significant advantages during labor. Being easily accessible, economical, and free of side effects, warm showers help relax muscles, improve circulation, reduce labor pain, and support a more positive maternal approach to the birth process. They ease fear and stress, promote comfort, and increase birth satisfaction. Studies indicate that pregnant women find warm showers soothing and often prefer them over analgesics. However, studies in Turkey on this subject are limited, and comprehensive research evaluating the combined effects of warm showers on labor pain, duration, emotional state, and breastfeeding is lacking. Therefore, this study was conducted to assess the effects of hydrotherapy during labor on these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women who were expected to give birth vaginally
* Women who became pregnant spontaneously
* Women who were in the latent phase of labor upon admission
* Women who were not given oxytocin
* Women who were at term (38-42 weeks of gestation)
* Women who had a single healthy fetus in the vertex position
* Women who did not have any risk factors (such as preeclampsia, eclampsia, placenta previa, or placental abruption).

Exclusion Criteria:

* Pregnant women with any complications that could cause dystocia during labor (such as contraction abnormalities birth objects, birth canal dystocia, maternal psychological dystocia)
* Who are unable to move
* Who cannot speak, read, or understand Turkish
* Who have communication problems.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | First time: Latent phase of labor, Second time: Second stage of labor (the stage in which the baby is born), Third time: Third stage of labor (the stage in which the placenta is born), Forth time: Second hour after birth
  The VAS is used to assess the pain felt. On the VAS, the patient marks the location of their pain on a ruler. This ruler is 10 cm long. One end of the ruler indicates no pain, and the other end indicates the most unbearable pain. The use of this scale must be explained very clearly to the pregnant woman. The pregnant woman is told that there are two endpoints on the ruler and that she should mark the point between these two endpoints that best represents the intensity of her pain. The distance between the "no pain" point and the point marked by the pregnant woman is measured in centimeters using the ruler and recorded. This determines the pregnant woman's pain level.
Breastfeeding Scoring System (LATCH) | Within the first two hours after birth
  The LATCH scale is a tool used to assess mothers' breastfeeding behaviors and skills. Developed by Jensen et al. in 1994, it evaluates five key areas: L (Latch onto the breast), A (Audible swallowing), T (Type of nipple), C (Comfort of breast/nipple), and H (Hold/positioning). Each criterion is scored 0 to 2 points, with a total score ranging from 0 to 10. Higher scores reflect more effective breastfeeding, while lower scores indicate potential difficulties. The scale's reliability and validity for the Turkish population were confirmed by Koyun (2001) and Okumuş and Yenal (2003). Widely used by healthcare professionals, the LATCH scale helps identify breastfeeding challenges early and supports mothers through education and intervention, promoting better breastfeeding outcomes and bonding.
Birth Emotion Scale (BES) | Within the first two hours after birth
  The Birth Emotion Scale (BES), developed by Hodnett in 1987, measures women's emotional experiences during childbirth. Gençalp validated and tested its reliability for the Turkish population in 1998. The scale contains 28 items scored on a 5-point Likert scale with options: "constantly," "frequently," "occasionally," "very rarely," and "never," coded from 1 to 5. Higher scores indicate more positive emotions during birth, while lower scores reflect negative emotions. Total scores range from 40 to 140. The Turkish version showed high internal consistency with a Cronbach's alpha of 0.87. The BES is widely used in research and clinical settings to assess psychological responses to childbirth and guide supportive care.
Labor Monitoring Form | First time: Latent phase of labor, Second time: Second stage of labor (the stage in which the baby is born), Third time: Third stage of labor (the stage in which the placenta is born), Forth time: Second hour after birth
  To determine labor stage durations in pregnant women, researchers recorded key time points during labor and delivery. These included hospital arrival, and transitions between labor stages: latent, active, transition phases, birth, placenta delivery, and transfer to the postpartum ward. Timing was measured in minutes for accuracy. The latent phase involves mild contractions and cervical dilation up to 4 cm. The active phase features stronger contractions and dilation from 4 to 7 cm. The transition phase completes dilation to 10 cm. Measuring these stages, along with placenta delivery and postpartum transfer, provides valuable data to assess labor progress, detect abnormalities, and evaluate interventions. This detailed timing supports improved obstetric care tailored to each woman's needs.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer Alan Dikmen, Assoc. Prof., Study Chair — Selcuk Uni̇versi̇ty
Locations (1):
- Mardin Eğitim ve Araştırma Hastanesi, Mardin, Midyat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomson G, Feeley C, Moran VH, Downe S, Oladapo OT. Women's experiences of pharmacological and non-pharmacological pain relief methods for labour and childbirth: a qualitative systematic review. Reprod Health. 2019 May 30;16(1):71. doi: 10.1186/s12978-019-0735-4. PMID 31146759
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Mallen-Perez L, Roe-Justiniano MT, Colome Ochoa N, Ferre Colomat A, Palacio M, Terre-Rull C. Use of hydrotherapy during labour: Assessment of pain, use of analgesia and neonatal safety. Enferm Clin (Engl Ed). 2018 Sep-Oct;28(5):309-315. doi: 10.1016/j.enfcli.2017.10.004. Epub 2017 Nov 24. English, Spanish. PMID 29239794
- [Background] M. (2018). "Comparing the effects of hot shower and intravenous injection of hyoscine on the pain intensity and duration of active phase of labour in nulliparous women". Journal of Clinical and Diagnostic Research, 12(8), QC07-QC11.
- [Background] Henrique AJ, Gabrielloni MC, Rodney P, Barbieri M. Non-pharmacological interventions during childbirth for pain relief, anxiety, and neuroendocrine stress parameters: A randomized controlled trial. Int J Nurs Pract. 2018 Jun;24(3):e12642. doi: 10.1111/ijn.12642. Epub 2018 Mar 7. PMID 29512230
- [Background] ACOG Committee Opinion No. 766: Approaches to Limit Intervention During Labor and Birth. Obstet Gynecol. 2019 Feb;133(2):e164-e173. doi: 10.1097/AOG.0000000000003074. PMID 30575638